CLINICAL TRIAL: NCT01638676
Title: A Phase I/II Trial of Vemurafenib and Metformin to Unresectable Stage IIIC and Stage IV BRAF.V600E+ Melanoma Patients
Brief Title: A Phase I/II Trial of Vemurafenib and Metformin to Melanoma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Chesney, Director, James Graham Brown Cancer Center, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-MEL-11-03
Record Dates: First submitted 2012-06-01; First posted 2012-07-12 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Melanoma
Keywords: Unresectable melanoma; Stage IIIC and Stage IV BRAFV600E+ Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib and Metformin (Experimental)
  Interventions: Drug: Vemurafenib; Drug: Metformin

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib (960 mg PO daily) in patients with unresectable BRAFV600E positive Stage IIIC and Stage IV melanoma
  Other Names: Vemurafenib branded as Zelboraf
Drug: Metformin — Metformin (500 mg PO BID x 2 weeks, then 850 mg PO BID)
  Other Names: Metformin hydrochloride branded as Glucophage

SUMMARY:
The main purpose of this study is to evaluate the safety of Vemurafenib in combination with Metformin in melanoma patients. The phase II part of the study will also evaluate the clinical activity of the combined regiment. Based on pre-clinical studies and a phase I trial, the investigators hypothesize that the combination of an FDA-approved non-toxic dose of oral Metformin with Vemurafenib will yield little toxicity and improve clinical outcomes in terms of objective response rates and survival in metastatic melanoma patients.

DETAILED DESCRIPTION:
This is a Phase I/II study. Phase I will be evaluating the safety of the FDA-approved Vemurafenib (960 mg orally, daily) in combination with Metformin (500 mg orally, twice daily for 2 weeks, then 850 mg orally,twice daily) in patients with unresectable Stage IIIC and Stage IV melanoma. Phase II will evaluate the clinical activity of the combined Vemurafenib/Metformin regimen. The safety profile of this combined Vemurafenib/Metformin regimen will be monitored during both phases. The treatment period consists of 28-day cycles until progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age;
2. Patients with histological confirmed BRAFV600E melanoma (Stage IIIC or Stage IV, American Joint Commission on Cancer);
3. Eastern Cooperative Oncology Group (ECOG) Performance Status(PS) of 0 to 2;
4. Life expectancy ≥ 3 months;
5. At least 1 site of radiographically measurable disease by RECIST 1.1
6. Adequate hematologic, renal, and liver function as defined by laboratory values performed within 42 days prior to initiation of dosing:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L;
   * Platelet count ≥ 50 x 109/L;
   * Hemoglobin ≥ 8 g/dL;
   * Serum creatinine ≤ 2 x upper limit of normal (ULN)
   * Total serum bilirubin ≤ 3 x ULN;
   * Serum aspartate transaminase (AST/SGOT) or serum alanine transaminase (ALT/SGPT) ≤ 3x ULN, and ≤ 4 x ULN if liver metastases are present.
7. Fertile males should use an effective method of contraception during treatment and for at least 3 months after completion of treatment, as directed by their physician;
8. Pre-menopausal females and females < 2 years after the onset of menopause should have a negative pregnancy test at Screening. Pre-menopausal females must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Females of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year;
9. Before study entry, written informed consent must be obtained from the patient prior to performing any study-related procedures.

Exclusion Criteria:

1. Prior treatment with Vemurafenib;
2. Known hypersensitivity to Metformin or any of its components;
3. Previous progression of melanoma while on Metformin;
4. Received radiotherapy for non CNS disease within the 2 weeks prior to commencing study treatment or have not recovered from side effects of all radiation-related toxicities to Grade ≤ 1, except for alopecia;
5. Pregnant, breast-feeding, or refusing double barrier contraception, oral contraceptives, or avoidance of pregnancy measures;
6. Have any other uncontrolled infection or medical condition that could interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Observation of CTCAE grade 4 or higher adverse events in six patients | Duration of phase I portion, approximately six months
  In the phase I portion, six patients will be enrolled and observed for CTCAE grade 4 or higher events. If three or more grade 4 or higher adverse events are observed among the six patients, the study will be halted.

SECONDARY OUTCOMES:
Overall Survival Follow up | Every 12 weeks (+/- 7 days) after last drug dose, for up to 3 full years
  Patients will be followed for up to three years following the last treatment administration. The Investigator or designees will make every possible attempt at least every 12 weeks (±7 days), for up to three years after the last treatment to contact the patient or family to obtain the survival information of the patient and, if applicable, the start date of additional anticancer treatment.
Number of adverse events | Duration of study, estimated to be approximately 60 months
  Descriptive statistics of all AEs observed during the study period.
type of adverse events | Duration of study, estimated to be approximately 60 months
  Descriptive statistics of all AEs observed during the study period.
Objective response rate (ORR)as measure of efficacy | Duration of study (approximately 60 months)
  Efficacy estimated as the objective response rate (ORR), which is the sum of Partial Responses (PR) and Complete Responses (CR) as determined by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Chesney, MD PhD, Principal Investigator — James Graham Brown Cancer Center-U of Louisville
Locations (1):
- James Graham Brown Cancer Center-University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Cerezo M, Tomic T, Ballotti R, Rocchi S. Is it time to test biguanide metformin in the treatment of melanoma? Pigment Cell Melanoma Res. 2015 Jan;28(1):8-20. doi: 10.1111/pcmr.12267. Epub 2014 Jun 26. PMID 24862830